CLINICAL TRIAL: NCT02722577
Title: Usefulness of Unipolar and Bipolar Electrograms in Predicting Successful Ablation Site During Idiopathic Outflow Tract Ventricular Arrhythmia Ablation
Brief Title: EGM Analysis in Idiopathic Outflow Tract Ventricular Arrhythmia
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: SJM-CIP-10090
Record Dates: First submitted 2016-03-08; First posted 2016-03-30 (Estimated); Results first posted 2019-07-29 (Actual); Last update posted 2019-08-06 (Actual); Status verified 2019-07

CONDITIONS: Ventricular Outflow Tract Tachycardia
MeSH Terms: interventions — Radiofrequency Ablation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Radio-frequency Ablation — A procedure that uses radiofrequency energy to destroy a small area of heart tissue that is causing rapid and irregular heartbeats.

SUMMARY:
Investigate the value of unipolar and bipolar electrograms (EGM) for predicting the successful ablation site for idiopathic outflow tract ventricular arrhythmia (OTVA).

DETAILED DESCRIPTION:
The proposed study aims to evaluate the predictive value of using reversed polarity in adjacent bipolar EGMs (bi-RP method) and unipolar EGM with QS morphology (uni-QS method) for identifying successful ablation site, and evaluate the feasibility of enhancing uni-QS method's performance by using its morphology characteristics such as descending slope and symmetry.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled to undergo ablation for idiopathic OTVA
* Have the ability to provide informed consent for study participation.

Exclusion Criteria:

* Be currently participating in any other investigational study
* Be less than 18 years of age
* Be pregnant
* Has any other conditions that are not suitable for catheter ablation (including but are not limited to active whole-body infection or sepsis, coagulation or hemorrhage disorder history)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 20 patients meeting the inclusion and exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guodong Niu, MD, Principal Investigator — Chinese Academy of Medical Sciences, Fuwai Hospital

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Presence of clinical arrhythmia during the ablation procedure is a requirement for the study protocol and can not be guaranteed at the time of enrollment. 2 of the patients who have consented did not have clinical arrhythmia present at the time of the ablation procedure and were therefore not included in the study.
Groups:
- Main Group: All patients enrolled in this study
Period: Overall Study
Arm/Group | Main Group
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Main Group
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 48 (16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 7
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  China | 20
Hypertension (%) [Count of Participants; unit: Participants] — Hypertension is measured in units of millimeters of mercury (mmHg). A subject is determined to have hypertension when the systolic blood pressure is higher than 130 mmHg or the diastolic blood pressure is higher than 80mmHg.
  Participants | 2
Diabetes mellitus (%) [Count of Participants; unit: Participants] — The diabetes mellitus condition is determined when the subject's Glycated hemoglobin level is 6.5 percent or higher on two separate tests.
  Participants | 0
Origin of arrhythmia in left ventricle outflow tract [Count of Participants; unit: Participants] — Determined when the subject's origin of arrhythmia was in left ventricle outflow tract during the electrocardiography testing.
  Participants | 4
QRS duration (ms) [Mean (Standard Deviation); unit: ms] | 147 (16)
Height (cm) [Mean (Standard Deviation); unit: cm] | 165 (8)
Weight (kg) [Mean (Standard Deviation); unit: kg] | 69 (9)

OUTCOME MEASURES:

1. Primary Outcome: Percent of Ablation Targets With Termination of the Clinical Ventricular Arrhythmia After RF Energy Delivery
Time Frame: Intraoperative, an average of 2 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Main Group
Number analyzed (Participants) | 20
Participants | 20

ADVERSE EVENTS:
Time Frame: Intraoperative, an average of 2 hours
Arm/Group | Main Group
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-03-01): https://cdn.clinicaltrials.gov/large-docs/77/NCT02722577/Prot_SAP_002.pdf